CLINICAL TRIAL: NCT03314064
Title: Long-term Safety of Subjects Continuing Dolutegravir After Participation in Clinical Studies of Dolutegravir in Russian Federation
Brief Title: Phase 4 Study of Dolutegravir (DTG) in Russian Federation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205908
Record Dates: First submitted 2017-10-13; First posted 2017-10-19 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: Phase 4; Russian Federation; dolutegravir; long-term safety; Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Intervention Model Description: This is an open label, single group study where the eligible subjects will receive DTG 50 mg once daily.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIV positive subjects continuing DTG (Experimental): HIV positive subjects who complete taking DTG in studies ING112276, ING113086, ING114915, ING111762 and those subjects who end participation in study 200304 in which they received either DTG or LPV/RTV will be included in this study.
  Interventions: Drug: Dolutegravir 50 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg — DTG is an integrase inhibitor that has been developed for ART of HIV-infection in combination with other antiretrovirals. DTG will be available as 50 mg tablets to be administered once daily.

SUMMARY:
DTG 50 milligram (mg) tablet was approved for marketing in Russian Federation; however, DTG is not currently available for subjects at Acquired Immune Deficiency Syndrome (AIDS) Centers as it is not available for order and supply via Federal program. This study is an open-label study which will include subjects, who complete taking DTG in studies ING112276, ING113086, ING114915, ING111762, and those subjects who end participation in study 200304 in which they received either DTG or lopinavir/ritonavir (LPV/RTV). DTG will be supplied at a dose of 50 mg once daily to eligible subjects until the subject stops taking DTG or transitions to commercial supply of DTG when available at AIDS Centers via the Federal program. The objective of this study is to bridge the gap between the closure of ING112276, ING113086, ING114915, ING111762 or end of subject's participation in 200304 and the actual availability of commercial DTG at AIDS Centers via Federal program for human immunodeficiency (HIV)-1-infected adult subjects in Russian Federation. The study will also investigate long-term safety of DTG for subjects continuing DTG in Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* The subject must complete an End of Study (EOS) visit for the originating protocol ING112276, ING113086, ING114915, ING111762, or be withdrawn from 200304 and attend withdrawal visit prior to transitioning to this study.
* Documented evidence of plasma HIV-1 RNA measurement <50 c/mL at the EOS visit in ING112276, ING113086, ING114915, ING111762, 200304 (for subjects receiving DTG ) and <400 c/mL for subjects prior receiving LPV/RTV in 200304.
* Based on medical assessment by the subject's Principal Investigator, the subject continues to derive clinical benefit from treatment with DTG as part of combination antiretroviral therapy (cART) and demonstrates stable virologic success. For subjects, currently receiving LPV/RTV and finishing their participation in 200304, possibility to derive clinical benefit from treatment with DTG is assessed by Principal Investigator following recommendation of Independent Data Monitoring Committee (IDMC).
* Subjects must be capable of giving signed informed consent to participate in this study.

Exclusion Criteria:

* Subjects not currently enrolled in clinical study ING112276, ING113086, ING114915, ING111762, 200304 are not eligible for this study.
* Subjects for whom confirmed virologic withdrawal criteria were met in ING112276, ING113086, ING114915, ING111762, 200304 are not eligible.
* In addition to the above mentioned criteria, investigator/physician must confirm that the subject has no prohibited clinical condition (other medicines or other health conditions, such as hepatic or renal contra-indications). Further, all women of child bearing potential must be cautioned that DTG is not approved for use in pregnancy, and be advised that birth control measures should be in place while taking DTG. Subjects who were permanently discontinued from DTG in the previous study due to intolerance must not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Number of subjects with drug related Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 7 months approximately
  Drug related AE is defined as all untoward and unintended responses to an investigational medicinal product related to any dose administered. All AEs will be graded according to Division of AIDS (DAIDS) toxicity scale.
Number of subjects with abnormal hematology parameters | Up to 7 months approximately
  Hematology parameters will be evaluated and will be graded according to DAIDS toxicity scale.
Number of subjects with abnormal clinical chemistry parameters | Up to 7 months approximately
  Clinical chemistry parameters will be evaluated and will be graded according to DAIDS toxicity scale.
Number of subjects with abnormal urine parameters | Up to 7 months approximately
  Urine parameters will be evaluated and will be graded according to DAIDS toxicity scale.
Number of subjects with abnormal electrocardiogram (ECG) | Up to 7 months approximately
  The number of subjects with abnormal ECG results will be summarized.
Number of subjects with abnormal radiological scan | Up to 7 months approximately
  The number of subjects with abnormal radiological scan will be summarized.
Number of subjects with abnormal physical examination | Up to 7 months approximately
  The number of subjects with abnormal physical examination will be summarized
Number of subjects with abnormal blood pressure | Up to 7 months approximately
  The number of subjects with abnormal blood pressure will be summarized.
Number of subjects with abnormal heart rate | Up to 7 months approximately
  The number of subjects with abnormal heart rate will be summarized.
Number of subjects with abnormal temperature | Up to 7 months approximately
  The number of subjects with abnormal body temperature will be summarized.
Number of subjects with abnormal respiratory rate | Up to 7 months approximately
  The number of subjects with abnormal respiratory rate will be summarized.
Number of subjects receiving concomitant medications | Up to 7 months approximately
  All the concomitant medications that the subject will receive will be evaluated.
Number of subjects achieving HIV-1 ribonucleic acid (RNA) suppression < 50 copies per milliliter (c/mL) | Up to 7 months approximately
  Efficacy of DTG will be assessed at routine clinical practice based on the maintenance of HIV-1 RNA suppression at <50 c/mL.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (10):
- Russia (10):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, N.Novgorod
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Toliyatti
  - GSK Investigational Site, Yekaterinburg